CLINICAL TRIAL: NCT03138850
Title: Comparison of Techniques to Improve Oxygenation and Capnographic Detection During Sedative Gastrointestinal Endoscopy
Brief Title: Improve Oxygenation and Capnographic Detection During Sedative EGD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-03-003B
Record Dates: First submitted 2017-04-18; First posted 2017-05-03 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-05

CONDITIONS: Upper Airway Obstruction; Apnea, Obstructive
Keywords: intravenous sedation; esophagogastroduodenalscopy; upper airway; mandibular advancement device; high flow nasal cannula
MeSH Terms: conditions — Airway Obstruction; Sleep Apnea, Obstructive | interventions — Cesarean Section

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Olympus standard bite block (Experimental): Standard of care using standard bite block and nasal cannula
  Interventions: Device: Olympus standard bite block
- YX Mandibular advancement bite block (Experimental): Mandibular advancement bite block group
  Interventions: Device: YX mandibular advancement bite block
- Optiflow High flow nasal cannula (Experimental): High flow nasal cannula group
  Interventions: Device: Optiflow High flow nasal cannula

INTERVENTIONS:
Device: Olympus standard bite block — Intravenous sedative upper gastrointestinal endoscopy performed under standard bite block (MB142 reusable bite block, Olympus) and nasal cannula with oxygen 5L/min
  Other Names: A
  Arms: Olympus standard bite block
Device: YX mandibular advancement bite block — Intravenous sedative upper gastrointestinal endoscopy performed under mandibular advancement bite block for endoscopy (Yong Xu breathing mouth piece, Yong Xu) and oxygen connected to mouth piece 5L/min
  Other Names: B
  Arms: YX Mandibular advancement bite block
Device: Optiflow High flow nasal cannula — Intravenous sedative upper gastrointestinal endoscopy performed under standard bite block (MB142 reusable bite block, Olympus) and high flow nasal cannula
  Other Names: C
  Arms: Optiflow High flow nasal cannula

SUMMARY:
The purpose of this study is to compare the effect of mandibular advancement bite block and high flow nasal cannula to standard bite block for oxygenation, capnographic measurement, prevention of hypoxemia, intervention events and adverse effects during endoscopic examinations.

DETAILED DESCRIPTION:
During endoscopic examinations, especially during those performed via oral insertion of endoscopes, an oral bite is used to protect the examination instruments and patients. During sedated endoscopic examinations, the patients are under influence of anesthetics. Upper airway obstruction often occurred due to respiratory depression and airway collapse resulting in desaturation. Airway management with high percentage oxygen, jaw thrust, or insertion of nasal airways by trained anesthetic personnel is required during upper airway obstruction emergencies. Nasal airway is invasive and causes nasal bleeding, sinusitis and other problems. Jaw thrust and bag-mask ventilation requires training and is a burden to anesthetic personnel to perform. Oxygenation and capnography are important ventilatory monitors during sedative procedures. These are often influenced by open mouth breathing during upper gastrointestinal endoscopic examinations making oxygenation and capnographic measurements unreliable. In this study, we group the patients into A group using standard of care, B group using mandibular advancement oral bite and C group using high-flow nasal cannulas. After anesthetic induction, gastric endoscopy will be performed. Oxygenation, end-tidal carbon dioxide, and degree of upper airway obstruction will be evaluated and recorded. Differences between the groups will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 20 to 80 years with ASA physical status I to II undergoing routine outpatient upper gastrointestinal endoscopy

Exclusion Criteria:

* Baseline oxygen saturation < 90%
* Known upper airway obstruction, difficult intubation history
* Unstable or lost of upper and lower incisors
* Known past oral or neck surgeries
* Anticipate exam time > 30 mins

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2017-06-22 (Actual); Study Completion 2017-06-22 (Actual)

PRIMARY OUTCOMES:
Area under the curve of 95% oxygen desaturation (AUCdesat) | From time of first sedative medication given until the time of discharge from recovery room, assessed up to 1 hour
  AUCdesat is defined as the integrated area under oxygen saturation (SPO2) for a selected cut point per 30 seconds, which better reflects the duration and severity of hypoxemia than the lowest saturation

SECONDARY OUTCOMES:
Number of rescue interventions | From time of first sedative medication given until the time of discharge from recovery room, assessed up to 1 hour
  Number of rescue interventions counted if any of the following procedures are performed, such as sustained chin lift or jaw thrust, insertion of an oral or nasal airway or bag-mask ventilation.
Number of apnea episodes | From time of first sedative medication given until the time of discharge from recovery room, assessed up to 1 hour
  Number of apnea episodes, which are number of times which the patient lack respiratory activity and loss of ETCO2 detection greater for 30 seconds occurs.
Number of partial airway obstruction episodes | From time of first sedative medication given until the time of discharge from recovery room, assessed up to 1 hour
  Number of partial airway obstruction episodes, which are number of times grunting or snoring with positive ETCO2 measurement greater than 30 secs occurs.
Number of total airway obstruction episodes | From time of first sedative medication given until the time of discharge from recovery room, assessed up to 1 hour
  Number of total airway obstruction episodes, which are number of times loss of ETCO2 detection while in presence of respiratory activity greater than 30 secs occurs.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Nung Teng, MD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Department of Anesthesiology, Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided